CLINICAL TRIAL: NCT04654832
Title: IVC Index in Patient With Diarrhea and Dehydration And How It Affects Its Management
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Refaat abd elhafez, Assistant lecturer, Assiut University
Other Study IDs: IVC Index
Record Dates: First submitted 2020-10-19; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Diarrhea, Infantile
Keywords: IVC Index
MeSH Terms: conditions — Diarrhea, Infantile

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
IVC Index in patient with Diarrhea and Dehydration And How It affects its management.

DETAILED DESCRIPTION:
Introduction The world health organization defines dehydration as condition that result from excessive loss of body water .the most common cause of dehydration in children are vomiting and diarrhea. Dehydration is a major cause of morbidity and mortality in infant and young children world wide .most cases due to consequence of acute gastroenteritis.

Pathophysiology. Dehydration cause decrease in total body water in both intracellular and extracellular fluid volume. Volume depletion closely correlate with sign and symptom of dehydration .the total body water is higher in infant and children compared to adult.

In infant, it is 70% of total body weight, whereas it is 65%and 60% respectively in children and adult.

The World Health Organization recommends assessing dehydration in children based on four clinical features: general appearance , eyes (whether they appear sunken), history of thirst , and skin pinch to assess turgor. However, these clinical signs may be subtle or non specific and thus have important limitations if used as independent predictors of dehydration. A more objective way to assess for dehydration using urine analysis has been implicated.

Additionally, studies on dehydration have shown urine analysis do not show sufficient sensitivity, Specificity or reliability [3, 4] and are typically only useful in children with moderate to severe hypovolemia.

. Bedside ultrasonography is a noninvasive method that can serve as a more objective tool for assessing dehydration in both adults and children. Point-of-care ultrasound has the potential to reduce unnecessary use of resources such as IV fluids or hospital access, while identifying children who are severely dehydrated and need immediate medical attention. Previous studies have shown that intravascular volume correlates to the diameters of the inferior vena cava.

* The normal IVC diameter is 15_ 17mm
* small IVC (usually < 12mm) with spontaneous collapse is often seen in the presence of intravascular volume depletion.

Bedside emergency ultrasonography (EUS) is a relatively new imaging modality in pediatrics.(8,9) EUS is fast, painless, and noninvasive. In recent years, many new pediatric indications for EUS have been developed.

Ultrasonography (US) assessment of the inferior vena cava (IVC) has been used as a noninvasive diagnostic tool for the assessment of intravascular volume and right heart function. Specifically, IVC diameter and collapsibility have been used as methods of assessing fluid status in dehydrated patients .

In these studies, contraction of the intravascular volume resulted in measurable decreases in IVC diameters. Conversely, research has shown that the diameter of the descending aorta (Ao) remains mostly constant, despite intravascular volume depletion.

ELIGIBILITY:
(Inclusion Criteria):

* Patients under 5years old who Presented with acute diarrhea and clinical evidence of significant (Moderate and severe) dehydration and sepsis based on blood picture ,high grade fever and CRP
* Patients under 5 years old with dehydration and non septic condition.
* Patients under 5years old have cardiomyopathy previously diagnosed.

(Exclusion Criteria ):

* Patients receiving oral rehydration solution only .
* chronic medical conditions, bronchopulmonary dysplasia and renal and liver diseases.
* Children with acute blood loss were also excluded.

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: *Sample size: According to the G*Power 3 software (Faul et al., 2007); the calculated minimum sample was 57 patient with dehydration needed to detect an effect size of 0.5 in the percentage of weight change after rehydration (12), with an error probability of 0.05 and 95 % power on a two-tailed test, it expected to be done from 1 October2020 till 29 December2021.(13)
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-29 (Estimated); Study Completion 2020-12-29 (Estimated)

PRIMARY OUTCOMES:
(IVC Index in patient with Diarrhea and Dehydration and how it affects it's management.) | IVC Index in patient with Diarrhea and Dehydration And How It affects its management21.(13). it expect it expected to be done from 1 October2020 till 29 December2021.(13)
  Assessment of dehydration by ivc index and bcmanagement according to this index

CONTACTS AND LOCATIONS:
Overall Officials: Elsayed Khalil Abd elkarem, Professor, Study Director — Assiut University; Duaa Mohamad raafat, Assistant, Study Director — Assiut University
Locations (1):
- Reham, Asyut, Egypt